CLINICAL TRIAL: NCT06582914
Title: Lynch Syndrome Integrative Epidemiology and Genetics (LINEAGE)
Brief Title: Lynch Syndrome Integrative Epidemiology and Genetics
Acronym: LINEAGE
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Chicago (Other); University of Kansas (Other); University of Pennsylvania (Other); Johns Hopkins University (Other); City of Hope National Medical Center (Other); Loma Linda University (Other); MedStar Health (Other); University of Arizona (Other); University of Manitoba (Other); University of Michigan (Other); University of North Carolina (Other); University of Pittsburgh (Other); University of Rochester (Other); Dana-Farber Cancer Institute (Other); University of Wisconsin, Madison (Other); The Cleveland Clinic (Other); University of California, San Diego (Other); Kaiser Permanente (Other); Ohio State University (Other); Virginia Mason Hospital/Medical Center (Other); University of Alabama at Birmingham (Other); University of Miami (Other)
Responsible Party: Sponsor
Other Study IDs: 24-0163
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Lynch Syndrome
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Years
Biospecimen Retention: Samples With DNA — A standardized procedure for collection and processing of human blood, stool, fresh frozen tissue, and formalin fixed paraffin embedded tissue for the LINEAGE Consortium can be used for all biosamples collected as part of the study. Barcoded samples will be stored at the clinical centers, using the specific labels for the LINEAGE study and corresponding data will be entered into the study database. Any center-specific processing differences should also be recorded by each center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pateints with a germline variant in a mismatch repair gene: Individuals with germline genetic testing results showing a pathogenic, likely pathogenic or variant of uncertain significance in MLH1, MSH2, MSH6, PMS2 or EPCAM.

SUMMARY:
The vision of the "Lynch syndrome INtegrative Epidemiology And GEnetics" (LINEAGE) Consortium is to collaboratively improve the lives and longevity of individuals and families with Lynch syndrome.

The mission of the LINEAGE Consortium is to collaboratively improve Lynch syndrome care through high-quality research. This consortium will provide intellectual and infrastructure support to facilitate development of research questions, collection of standardized data and biospecimens, support of grant applications, and generation of collaborative manuscripts.

Our aims are to:

I. Establish a prospective cohort of individuals with Lynch syndrome II. Collect standardized longitudinal clinical and biosample data to elucidate Lynch Syndrome epidemiology and gene-host interactions III. Promote intervention trials to improve cancer prevention and early detection in Lynch Syndrome

DETAILED DESCRIPTION:
The main objective of this consortium is to build a shared resource to drive research in critical areas necessary to understand LS-related neoplasia risk and improve early detection and prevention of LS-associated cancers. This consortium will provide intellectual and infrastructure support to facilitate development of research questions, collection of standardized clinical data and biospecimens, support grant applications, and generate collaborative manuscripts.

Data and samples collected for LINEAGE will allow the consortium to address a variety of topic areas including but not limited to:

I. Risk of prevalent and incident colorectal neoplasia among PV/LPV carriers. II. Estimate risk of prevalent and incident extra-colonic neoplasm among PV/LPV carriers.

III. Characterization of post-colonoscopy colorectal cancer among PV/LPV carriers.

IV. Risk factors for prevalent and incident neoplasia.

The LINEAGE Consortium is an observational prospective cohort study, with baseline and annual electronic health record (EHR) abstraction, and electronic participant and provider surveys. The consortium may also collect single or serial biosamples from identified and enrolled LS patients at participating centers.

ELIGIBILITY:
Inclusion Criteria:

* • Adults age over 18 years

  * Eligible patients must have at least one variant of uncertain significance (VUS), pathogenic or likely pathogenic variant (PV/LPV) in MLH1, MSH2, MSH6, PMS2, or EPCAM, which will be confirmed by genetic testing results (obtained as part of routine care) and a review of the variant in ClinVar (https://www.ncbi.nlm.nih.gov/clinvar/).
  * Individuals who are an obligate carrier of a LS PV/LPV that is confirmed in the family.

Exclusion Criteria:

* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Lynch Syndrome, defined as having a pathogenic or likely pathogenic variant in a mismatch repair gene (MLH1, MSH2, MSH6, PMS2, EPCAM) on germline genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2054-12-31 (Estimated); Study Completion 2054-12-31 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer incidence | 40 years
  cases of adenocarcinoma of the colon or rectum diagnosed over the observation period

SECONDARY OUTCOMES:
non-colorectal cancer incidence | 40 years
  new cases of any cancer diagnosed over observation period
precancerous colorectal polyps | 40 years
  new diagnoses of any of the following polyps in the colon or rectum
  * tubular adenoma
  * villous adenoma
  * tubulovillous adenoma
  * sessile serrated lesion
  * traditional serrated adenoma

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado, Aurora, Colorado
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No
We do not have IRB approval to do this at this time.

REFERENCES:
- [Background] Yao MD, von Rosenvinge EC, Groden C, Mannon PJ. Multiple endoscopic biopsies in research subjects: safety results from a National Institutes of Health series. Gastrointest Endosc. 2009 Apr;69(4):906-10. doi: 10.1016/j.gie.2008.05.015. Epub 2009 Jan 10. PMID 19136110
- [Background] Kind AJH, Buckingham WR. Making Neighborhood-Disadvantage Metrics Accessible - The Neighborhood Atlas. N Engl J Med. 2018 Jun 28;378(26):2456-2458. doi: 10.1056/NEJMp1802313. No abstract available. PMID 29949490
- [Background] Dominguez-Valentin M, Sampson JR, Seppala TT, Ten Broeke SW, Plazzer JP, Nakken S, Engel C, Aretz S, Jenkins MA, Sunde L, Bernstein I, Capella G, Balaguer F, Thomas H, Evans DG, Burn J, Greenblatt M, Hovig E, de Vos Tot Nederveen Cappel WH, Sijmons RH, Bertario L, Tibiletti MG, Cavestro GM, Lindblom A, Della Valle A, Lopez-Kostner F, Gluck N, Katz LH, Heinimann K, Vaccaro CA, Buttner R, Gorgens H, Holinski-Feder E, Morak M, Holzapfel S, Huneburg R, Knebel Doeberitz MV, Loeffler M, Rahner N, Schackert HK, Steinke-Lange V, Schmiegel W, Vangala D, Pylvanainen K, Renkonen-Sinisalo L, Hopper JL, Win AK, Haile RW, Lindor NM, Gallinger S, Le Marchand L, Newcomb PA, Figueiredo JC, Thibodeau SN, Wadt K, Therkildsen C, Okkels H, Ketabi Z, Moreira L, Sanchez A, Serra-Burriel M, Pineda M, Navarro M, Blanco I, Green K, Lalloo F, Crosbie EJ, Hill J, Denton OG, Frayling IM, Rodland EA, Vasen H, Mints M, Neffa F, Esperon P, Alvarez K, Kariv R, Rosner G, Pinero TA, Gonzalez ML, Kalfayan P, Tjandra D, Winship IM, Macrae F, Moslein G, Mecklin JP, Nielsen M, Moller P. Cancer risks by gene, age, and gender in 6350 carriers of pathogenic mismatch repair variants: findings from the Prospective Lynch Syndrome Database. Genet Med. 2020 Jan;22(1):15-25. doi: 10.1038/s41436-019-0596-9. Epub 2019 Jul 24. PMID 31337882
- [Background] Win AK, Jenkins MA, Dowty JG, Antoniou AC, Lee A, Giles GG, Buchanan DD, Clendenning M, Rosty C, Ahnen DJ, Thibodeau SN, Casey G, Gallinger S, Le Marchand L, Haile RW, Potter JD, Zheng Y, Lindor NM, Newcomb PA, Hopper JL, MacInnis RJ. Prevalence and Penetrance of Major Genes and Polygenes for Colorectal Cancer. Cancer Epidemiol Biomarkers Prev. 2017 Mar;26(3):404-412. doi: 10.1158/1055-9965.EPI-16-0693. Epub 2016 Oct 31. PMID 27799157